CLINICAL TRIAL: NCT07139678
Title: Turkish Reliability and Validity of the Safe Use of Mobility Aids Checklist (SUMAC) For 4-wheeled Walker Use
Brief Title: Safe Use of Mobility Aids Checklist (SUMAC) for 4-wheeled Walker Use in Turkish Geriatric Population
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1173
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: dependent ambulation; dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric participants: Participants with dementia who are 65 years old or older
  Interventions: Other: SUMAC

INTERVENTIONS:
Other: SUMAC — Participant will complete tasks given in SUMAC.

SUMMARY:
The goal of this observational study is to investigate the validity and reliability of the Safe Use of Mobility Aids Checklist (SUMAC) for 4-wheeled walker use in Turkish geriatric population. The main questions it aims to answer are:

Is SUMAC reliable for Turkish geriatric population? Is SUMAC valid for Turkish geriatric population?

Participants will fill out questionnaires and perform the tasks given in SUMAC.

DETAILED DESCRIPTION:
Participants with dementia who are older than 65 years will be evaluated through some questionnaires such as Katz Index of Independence in Activities of Daily Living (ADL) and Mini-Mental State Examination. They will perform the Tinetti Test and their walking speed will also be measured. Participants will perform 9 tasks stated in SUMAC and will be recorded so that the investigators can score the tasks.

Tasks include: Transition of Sit to Stand, Gait with Pivot Turn To Approach Chair To Sit, Ambulation on a Level Surface, Walking While Performing Task of Horizontal Head Turns, Walking While Performing a Concurrent Cognitive Task, Walking While Negotiating Obstacles, Walking Through an Open Doorway, Open and Walk Through a Door that Opens Away From Person, Open and Walk Through Door that Opens Towards the Person.

This study contains 4 phases. Firstly, SUMAC will be translated to Turkish by two people whose native language is Turkish and who have full knowledge of the test terminology along with advanced knowledge of English. The Turkish version will be back translated to English by two native English speakers who are not connected to this study. The final translation will be determined by the committee which includes four translators and one Turkish philologist. In the second phase, participants will be filmed during their performances of the nine tasks in SUMAC. For recording, permission will be attained from participants and the people who are in charge of their care.

Recordings will be kept in a computer protected by a password, and will be deleted once the study is completed. For the third phase, a team of physiotherapists will complete the training for every taks in SUMAC in order to evaluate participants. In the fourth phase, SUMAC's reliability and validity for a Turkish geriatric population with dementia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosed dementia
* Using 4-wheeled walker
* Being 65 years old or older
* Being able to understand and speak Turkish
* Having graduated from at least middle school
* Being able to follow the instructions and act accordingly
* Being able to walk without another person's help
* Having gotten 18-23 points from the The Mini Mental State Examination (MMSE)

Exclusion Criteria:

* Having mobility limitations due to musculoskeletal and neurological problems
* Having problems walking due to neurological diseases such as Parkinson, cerebrovascular diseases and so on
* Having balance problems due to vestibular conditions
* Having severe visual impairment and/or severe hearing loss
* Having unstable cardiovascular diseases
* Having malignancy and/or receiving treatment for malignancy
* Having had a surgery related to neurological and/or orthopedic problems in the past 6 months
* Not being willing to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People who are 65 years or older with dementia will be included in the study. Participants will be selected from nursing homes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
The Safe Use of Mobility Aids Checklist (SUMAC) for 4-wheeled walker | 7 days
  Participants will perform the tasks given in SUMAC. For reliability, they will perform the same tasks one week later.

SECONDARY OUTCOMES:
The Tinetti Test | 15 days
  The scores of the test will be used to determine the validity of Turkish SUMAC.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Kaya, RA, Study Director — Ankara Yildirim Beyazıt University; Bahar Anaforoğlu, Prof., Principal Investigator — Ankara Yildirim Beyazıt University; Nezehat Ö Ünlüer, Assoc. Prof., Study Director — Saglik Bilimleri Universitesi; Yasemin Ateş Sarı, Dr., Study Director — Ankara Yildirim Beyazıt University; Büşra Kalkan Balak, TA, Study Director — Yüksek İhtisas University; Sevilay S Baş, Dr., Study Director — Ankara Yildirim Beyazıt University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrer A, Formiga F, Sanz H, de Vries OJ, Badia T, Pujol R; OCTABAIX Study Group. Multifactorial assessment and targeted intervention to reduce falls among the oldest-old: a randomized controlled trial. Clin Interv Aging. 2014 Feb 25;9:383-93. doi: 10.2147/CIA.S57580. eCollection 2014. PMID 24596458
- [Background] Shumway-Cook A, Ciol MA, Hoffman J, Dudgeon BJ, Yorkston K, Chan L. Falls in the Medicare population: incidence, associated factors, and impact on health care. Phys Ther. 2009 Apr;89(4):324-32. doi: 10.2522/ptj.20070107. Epub 2009 Feb 19. PMID 19228831
- [Background] Hartholt KA, van Beeck EF, Polinder S, van der Velde N, van Lieshout EM, Panneman MJ, van der Cammen TJ, Patka P. Societal consequences of falls in the older population: injuries, healthcare costs, and long-term reduced quality of life. J Trauma. 2011 Sep;71(3):748-53. doi: 10.1097/TA.0b013e3181f6f5e5. PMID 21045738
- [Background] Tan MP, Kamaruzzaman SB, Zakaria MI, Chin AV, Poi PJ. Ten-year mortality in older patients attending the emergency department after a fall. Geriatr Gerontol Int. 2016 Jan;16(1):111-7. doi: 10.1111/ggi.12446. Epub 2015 Jan 22. PMID 25613422
- [Background] Frith, K. H., Hunter, A. N., Coffey, S. S., & Khan, Z. (2019). A longitudinal fall prevention study for older adults. The journal for nurse practitioners, 15(4), 295-300.
- [Background] Bateni H, Maki BE. Assistive devices for balance and mobility: benefits, demands, and adverse consequences. Arch Phys Med Rehabil. 2005 Jan;86(1):134-45. doi: 10.1016/j.apmr.2004.04.023. PMID 15641004
- [Background] Hartke RJ, Prohaska TR, Furner SE. Older adults and assistive devices: use, multiple-device use, and need. J Aging Health. 1998 Feb;10(1):99-116. doi: 10.1177/089826439801000106. PMID 10182420
- [Background] Hardi I, Bridenbaugh SA, Gschwind YJ, Kressig RW. The effect of three different types of walking aids on spatio-temporal gait parameters in community-dwelling older adults. Aging Clin Exp Res. 2014 Apr;26(2):221-8. doi: 10.1007/s40520-014-0204-4. Epub 2014 Mar 12. PMID 24619887
- [Background] Resnik L, Allen S, Isenstadt D, Wasserman M, Iezzoni L. Perspectives on use of mobility aids in a diverse population of seniors: implications for intervention. Disabil Health J. 2009 Apr;2(2):77-85. doi: 10.1016/j.dhjo.2008.12.002. PMID 20160951
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Liu HH. Assessment of rolling walkers used by older adults in senior-living communities. Geriatr Gerontol Int. 2009 Jun;9(2):124-30. doi: 10.1111/j.1447-0594.2008.00497.x. PMID 19740354
- [Background] Liu HH, Eaves J, Wang W, Womack J, Bullock P. Assessment of canes used by older adults in senior living communities. Arch Gerontol Geriatr. 2011 May-Jun;52(3):299-303. doi: 10.1016/j.archger.2010.04.003. Epub 2010 Apr 22. PMID 20416960
- [Background] Hunter SW, Omana H, Madou E, Wittich W, Hill KD, Johnson AM, Divine A, Holmes JD. Effect of dual-tasking on walking and cognitive demands in adults with Alzheimer's dementia experienced in using a 4-wheeled walker. Gait Posture. 2020 Mar;77:164-170. doi: 10.1016/j.gaitpost.2020.01.024. Epub 2020 Feb 1. PMID 32044696
- [Background] Hunter SW, Divine A, Omana H, Wittich W, Hill KD, Johnson AM, Holmes JD. Effect of Learning to Use a Mobility Aid on Gait and Cognitive Demands in People with Mild to Moderate Alzheimer's Disease: Part II - 4-Wheeled Walker. J Alzheimers Dis. 2019;71(s1):S115-S124. doi: 10.3233/JAD-181170. PMID 31127767
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Arik G, Varan HD, Yavuz BB, Karabulut E, Kara O, Kilic MK, Kizilarslanoglu MC, Sumer F, Kuyumcu ME, Yesil Y, Halil M, Cankurtaran M. Validation of Katz index of independence in activities of daily living in Turkish older adults. Arch Gerontol Geriatr. 2015 Nov-Dec;61(3):344-50. doi: 10.1016/j.archger.2015.08.019. Epub 2015 Aug 28. PMID 26328478
- [Background] Shubert TE, Schrodt LA, Mercer VS, Busby-Whitehead J, Giuliani CA. Are scores on balance screening tests associated with mobility in older adults? J Geriatr Phys Ther. 2006;29(1):35-9. PMID 16630375
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Hunter SW, Divine A, Omana H, Madou E, Holmes J. Development, reliability and validity of the Safe Use of Mobility Aids Checklist (SUMAC) for 4-wheeled walker use in people living with dementia. BMC Geriatr. 2020 Nov 11;20(1):468. doi: 10.1186/s12877-020-01865-5. PMID 33176695
- [Background] Yücel, S. D., Şahin, F., Doğu, B., Şahin, T., Kuran, B., & Gürsakal, S. (2012). Reliability and validity of the Turkish version of the Performance-Oriented Mobility Assessment I. European Review of Aging and Physical Activity, 9(2), 149-159.
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Safe Use of Mobility Aids Checklist (SUMAC) documents (2022, October 25), retrieved from: http://www.mobility-in-aging-lab.ca/#publications